CLINICAL TRIAL: NCT04440813
Title: The Risk of HIV Acquisition Among Traditional Healers in South Africa: Implementing Novel Strategies to Improve Protective Behaviors
Brief Title: The Risk of HIV Acquisition Among Traditional Healers in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Carolyn Audet, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21AI150302 (NIH); R21AI150302-01 (NIH)
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician Training (Active Comparator): Traditional healers randomized to the control arm will receive PPE education and training, general HIV prevention education and skill building (including condom use, positive prevention, and pre-/post-exposure prophylaxis services), and three educational outreach and coaching visits at the healer's place of practice to provide on-the-ground advice and support for PPE use. All training will be provided by trained medical personnel.
  Interventions: Behavioral: Education and Training by Clinicians
- Healer + Clinician Training (Experimental): Traditional healers randomized to the intervention arm will receive PPE education and training, general HIV prevention education and skill building (including condom use, positive prevention, and pre-/post-exposure prophylaxis services), and three educational outreach and coaching visits at the healer's place of practice to provide on-the-ground advice and support for PPE use. All training will be provided by both healers who already use PPE regularly and trained medical personnel.
  Interventions: Behavioral: Training and Education from Traditional Healers and Clinicians

INTERVENTIONS:
Behavioral: Education and Training by Clinicians — Training in the use of PPE and education about the risks of blood exposure.
  Arms: Clinician Training
Behavioral: Training and Education from Traditional Healers and Clinicians — Training in the use of PPE and education about the risks of blood exposure.
  Arms: Healer + Clinician Training

SUMMARY:
Traditional healers, community-based partners with the national health system of South Africa, are exposed to patient blood an average of 1,500 times during their careers due to the practice of delivering herbal remedies via herbs rubbed into dozens of sub-cutaneous cuts. The purpose of this proposal is to compare two implementation strategies to increase consistent use of Personal Protective Equipment (PPE): (1) a health care worker provided training program followed by 3 educational outreach and coaching visits at the healer's place of practice vs. (2) a training and educational outreach initiative led by a team of health care workers and healers who adopted and use PPE on their own (early adopters) to assess their effects on exposure to patient blood. With an HIV prevalence among healers well above that in the baseline population (30% vs. 19%) and HIV prevalence of 59% among those exposed to patient blood, this study will allow the investigators to test a novel implementation strategy for delivering PPE training to prevent new HIV infections among a newly identified high-risk population in a region with the world's highest HIV prevalence.

DETAILED DESCRIPTION:
In South Africa there are an estimated 200,000 traditional healers providing health services. Like allopathic health care workers (HCW), traditional healers are exposed to bloodborne pathogens through the widespread practice of traditional "injections", where healers perform dozens of subcutaneous incisions to rub herbs directly into the bloodied skin. 98 percent of healers perform these treatments; they experience an average of 1,500 blood exposures over the course of their lifetime. This high frequency of blood exposure, coupled with treating high-risk patients, can result in an increased risk of patient-to-healer disease transmission if personal protective equipment (PPE) are not used. Healers in South Africa who reported patient blood touched their skin had 2.59 times higher risk of being HIV-positive than those with no exposure (59% vs. 25%); overall healers have a substantially higher HIV prevalence (30%) than the general population (19%).

Free PPE are made available at local health facilities, but most healers have low levels of literacy, limited ability to assess blood exposure risk, and have no PPE training. Given these limitations, use of PPE during treatments is inconsistent. A small proportion of healers employ PPE appropriately during each treatment; these "early adopter" healers suggest PPE use is sustainable in rural sub-Saharan Africa if a healer has the necessary skills, risk assessment training, and encouragement. This proposal compares two implementation strategies to increase PPE use during procedures and decrease the number of injections performed: (1) HCW led education on risk of blood exposure and development of PPE donning, use and doffing skills through a week-long training followed by 3 educational outreach visits at the healer's place of practice vs. (2) "Early adopter" healer and HCW co-led week-long training followed by 3 educational outreach visits. The investigators hypothesize that the strategy of engaging "early adopter" healers as trainers will lead to more accurate participant risk assessments, increase participant self-efficacy, and lead to more consistent use of PPE during treatments.

The Specific Aims of this study are to:

1. Adapt PPE training using the "ADAPT-ITT" model;
2. Compare fidelity of PPE training between the HCW-only team versus the healer + HCW team;
3. Compare the effects of two implementation strategies on healer exposure to patient blood.

This potentially high-impact intervention is well-suited to the R21 mechanism. While some allopathic providers may recommend an outright ban on the procedure, patients and healers have strongly believed in the efficacy of these treatments for hundreds of years- they are not likely to stop because of a Department of Health recommendation. It is up healthcare workers and governments to overcome their own biases to develop an effective strategy to prevent HIV seroconversion. The team of South African and U.S. investigators has a proven record of HIV research success and specific experience successfully engaging traditional healers, HIV prevention studies, as well as, dissemination and implementation research.

ELIGIBILITY:
Inclusion Criteria:

1. Traditional healers > 18 years of age, who are registered as traditional healers with the government of South Africa, are currently practicing in the Bushbuckridge area, and conduct traditional vaccinations.
2. Biomedical practitioners > 18 years of age, who are currently providing health care services to patients at government or private health facilities in Bushbuckridge. '
3. Community members > 18 years of age, who currently live in Bushbuckridge and sought health care services from a traditional healer in the past year.

Exclusion Criteria:

1. Traditional healers <18 years of age, who are not registered as traditional healers with the government of South Africa, are not currently practicing, or do not conduct traditional vaccinations on their patients.
2. Biomedical practitioners < 18 years of age or who are not currently providing health services in the Bushbuckridge area.
3. Community members < 18 years of age or who do not seek health care services from traditional healers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn M Audet, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Ludlow, Ludlow, MPM, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Audet CM, Seabi T, Oyekunle T, Hove J, Wagner RG. A individually randomized controlled trial comparing Healer-led vs. clinician- led training to improve personal protective equipment use among traditional healers in South Africa. PLOS Glob Public Health. 2024 Feb 23;4(2):e0002945. doi: 10.1371/journal.pgph.0002945. eCollection 2024. PMID 38394119

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinician Training | Healer + Clinician Training
Started | 69 | 67
Completed | 64 | 62
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinician Training | Healer + Clinician Training | Total
Number analyzed (Participants) | 69 | 67 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (12.64) | 53 (14.18) | 51.0 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 53 | 110
  Male | 12 | 14 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 69 | 67 | 136
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 69 | 67 | 136
HIV knowledge- HIV is caused by curse [Count of Participants; unit: Participants]
  Answered correctly | 42 | 38 | 80
  Answered incorrectly | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Blood Exposure
Description: Number of Glove Pairs Used Per Razor Blade Used
Time Frame: 7 months
Population: Some of the traditional healers did not conduct any traditional vaccinations during the study period, thus our numbers are smaller than the total number of participants
Measure: Mean (Standard Deviation); unit: Number of Glove Pairs Used Per Razor Bla
Arm/Group | Clinician Training | Healer + Clinician Training
Number analyzed (Participants) | 53 | 60
Number of Glove Pairs Used Per Razor Bla | 1.9 (0.79) | 1.9 (0.73)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Clinician Training | Healer + Clinician Training
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/67
Other Adverse Events (participants affected / at risk) | 0/69 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT04440813/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT04440813/ICF_001.pdf